CLINICAL TRIAL: NCT01375140
Title: Evaluation of Ruxolitinib and Lenalidomide Combination as a Therapy for Patients With Myelofibrosis
Brief Title: Ruxolitinib and Lenalidomide for Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0269; NCI-2011-01126 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-06-14; First posted 2011-06-17 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Myeloproliferative Diseases
Keywords: Myeloproliferative Diseases; Myelofibrosis; Post essential thrombocythemia/polycythemia vera; Ruxolitinib; INCB018424; Lenalidomide; CC-5013; Revlimid; Prednisone; Interactive Voice Response System; IVR
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera | interventions — ruxolitinib; Lenalidomide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib + Lenalidomide (Experimental): Ruxolitinib 15 mg orally twice daily continuously + Lenalidomide orally 5 mg/day on days 1-21, followed by 7 days of no therapy (28-day cycle). Prednisone will be added for patients who have not responded after 3 cycles of therapy. Prednisone 30 mg by mouth a day during cycle 4, 15 mg/day during cycle 5, and 15 mg every other day during cycle 6, and then it will be discontinued.
  Interventions: Drug: Ruxolitinib; Drug: Lenalidomide; Drug: Prednisone

INTERVENTIONS:
Drug: Ruxolitinib — 15 mg by mouth twice daily (BID), continuously in 28-day cycles.
  Other Names: INCB018424
Drug: Lenalidomide — 5 mg by mouth each day on days 1-21, followed by 7 days of no therapy of each 28 day cycle.
  Other Names: CC-5013; Revlimid
Drug: Prednisone — Prednisone will be added for patients who have not responded after 3 cycles of therapy.
  30 mg by mouth a day during cycle 4, 15 mg/day during cycle 5, and 15 mg every other day during cycle 6, and then it will be discontinued.

SUMMARY:
The goal of this clinical research study is to learn if the combination of ruxolitinib and lenalidomide can help to control MF. The safety of this study drug combination will also be studied.

Ruxolitinib is designed to stop certain proteins (called JAK1 and JAK2) that are found in MF cells from sending signals that may lead to the growth of cancer cells.

Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. This may decrease the growth of cancer cells.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found eligible to take part in this study, you will begin taking ruxolitinib by mouth 2 times every day during each 28-day cycle. You should take ruxolitinib one time in the morning and one time in the evening (about 12 hours apart). Ruxolitinib should be taken with a meal and a glass of water. If you miss a dose of ruxolitinib, you should not make up the dose or take any more before the next scheduled dose.

You will also take lenalidomide by mouth one time in the morning on Days 1-21 of each cycle. Lenalidomide capsules should be swallowed whole, and should not be broken, chewed, or opened. If a dose of lenalidomide is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should not be made up.

If your study doctor thinks it is needed or if you have side effects, your dose of ruxolitinib and/or lenalidomide may be stopped, lowered, or delayed for up to 8 weeks during the study.

During the study, you will need to return all unused study drug to the study staff at each clinic visit.

Additional Drugs:

If your disease has not responded to the study drugs after 3 cycles and the study doctor thinks it is in your best interest, you may begin taking prednisone along with the study drugs. Prednisone is a corticosteroid that is similar to a natural hormone made by your body. Prednisone is often given in combination with other chemotherapy drugs. You will take prednisone every morning during Cycles 4 and 5, then every other day during Cycle 6. After Cycle 6, you will no longer take prednisone. If you forget to take a does of prednisone and more than 8 hours have passed, wait until the next day to take prednisone again (or 2 days later if you are taking it every other day during Cycle 6).

If your doctor thinks it is needed, you may take aspirin during this study to help prevent blood clots from forming. If you are allergic to aspirin or cannot take aspirin, your doctor may recommend you take another type of drug to help prevent blood clots from forming.

Study Drug Diary:

You will be given a study drug diary before you begin taking the study drugs to write down what time you take each dose of the study drugs. You will need to bring the diary with you to each study visit so it can be reviewed.

You should bring the study drug (including empty bottles) with you to all of the study visits. You will be asked not to take your morning dose of study drug before your visits on Day 15 Cycle 1 and Day 1 on Cycle 2.

Study Visits:

On Day 1 of Cycles 1 and 2:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Blood (about 3 teaspoons) will be drawn for routine tests and to check your kidney and liver function. This routine blood draw will include a pregnancy test if you are able to become pregnant.
* You will complete 2 questionnaires about your quality of life. The questionnaires should take about 10 minutes to complete. One of the questionnaires may be filled out on a computer. The study staff will help you use the computer.

On Days 8 and 22 of Cycles 1 and 2:

° Blood (about 3 teaspoons) will be drawn for routine tests. This routine blood draw will include a pregnancy test if you are able to become pregnant.

On Day 15 of Cycles 1 and 2:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any side effects you may be having.
* Blood (about 3 teaspoons) will be drawn for routine tests and to check your kidney and liver function. This routine blood draw will include a pregnancy test if you are able to become pregnant.

On Day 1 of Cycle 3 and every 3 to 6 Cycles after that:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a review of any blood transfusions you may have had in the last 3 months.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Blood (about 3 teaspoons) will be drawn for routine tests and to check your kidney and liver function. This routine blood draw will include a pregnancy test if you are able to become pregnant.
* You will complete 2 questionnaires about your quality of life. The questionnaires should take about 10 minutes to complete.

You will have a bone marrow biopsy and aspirate after Cycles 3, 6, 9, and 12, and then when your doctor feels it is necessary.

Interactive Voice Response (IVR) System:

During the first 3 cycles, you will use the Interactive Voice Response (IVR) system once a month to tell the study staff about any side effects you may be having. The IVR system is an automated calling system that will allow you to press buttons on your phone to answer questions about any side effects you may be having. The study staff will give you instructions on how to use the IVR. If you are not able to use the IVR system, a member of the study staff will contact you instead.

After Cycle 3, a member of the study staff will call you at your home once a month to ask you about any side effects you may be having and to review the results of your blood tests.

Length of Study:

You may receive the study drug combination for up to 6 years. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

You will be considered off study after your follow-up visit.

End-of-Study Visit:

You will have an end-of-study visit the day you are taken off study. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a review of any blood transfusions you may have had in the last 3 months.
* You will be asked about any drugs you may be taking and any side effects you may be having.
* Blood (about 3 teaspoons) will be drawn for routine tests and to check your kidney and liver function. This routine blood draw will include a pregnancy test if you are able to become pregnant.
* You will complete 2 questionnaires about your quality of life. The questionnaires should take about 10 minutes to complete.
* You will have a bone marrow biopsy and/or aspirate to check the status of the disease.

Follow-up:

A member of the study staff will call you 30 days and 60 days after you have stopped taking the study drugs to ask how you are feeling and if you have had any side effects since your last visit.

This is an investigational study. Lenalidomide is not FDA-approved or commercially available for use in patients with MF. Ruxolitinib is FDA approved and commercially available for the treatment of intermediate or high-risk myelofibrosis, including primary myelofibrosis, post-polycythemia vera (post-PV) myelofibrosis and post-essential thrombocythemia (post-ET) myelofibrosis. Lenalidomide is FDA-approved for the treatment of some forms of myelodysplastic syndrome (MDS) and multiple myeloma (MM). Its use in patients with MF is investigational.

Up to 49 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of myelofibrosis (either primary or post essential thrombocythemia/polycythemia vera) requiring therapy, including those previously treated and relapsed or refractory, or if newly diagnosed, with intermediate-1 or -2 or high risk according to International Working Group (IWG) criteria.
2. Understanding and voluntary signing an IRB-approved informed consent form.
3. Age equal to or greater than 18 years at the time of signing the informed consent.
4. Disease-free of prior malignancies for equal to or greater than 2 years with exception of basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
5. ECOG performance status 0 to 2.
6. Patients must have adequate organ function as demonstrated by the following: a. Direct bilirubin equal to or less than 2.0 mg/dL, b. Serum creatinine equal to or less than 2.0 mg/dL., c. SGPT equal to or less than 3 x upper limit of normal
7. Females of childbearing potential (FCBP)(A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
8. Cont. from 7: must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 to 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
9. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
10. Platelets >/= 100000/uL
11. ANC >/= 1000/uL

Exclusion Criteria:

1. Use of any other standard (e.g. hydroxyurea, anagrelide, growth factors) or experimental drug or therapy within 14 days or 5-half lives, whichever is longer, of starting study therapy and/or lack of recovery from all toxicity from previous therapy to grade 1 or better.
2. Known prior clinically relevant hypersensitivity reaction to thalidomide, including the development of erythema nodosum if characterized by a desquamating rash.
3. Prior therapy with lenalidomide or ruxolitinib.
4. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
5. Suspected Pregnancy, Pregnant or lactating females.
6. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
7. Known positive for HIV or infectious hepatitis, type A, B or C.
8. Known prior clinically relevant hypersensitivity to prednisone.
9. Participants with prior history of thromboembolic disease (i.e. deep venous thrombosis (DVT) or pulmonary embolism (PE) within the last six months, as Lenalidomide has demonstrated a significantly increased risk of DVT or PE.
10. Known to have a hypercoagulability syndrome (eg: antithrombin III, deficiency, anticardiolipin syndrome etc…)
11. Concurrent use of strong inducers or strong inhibitors of CYP3A4 (strong inducers are rifampin and St. John's Worth, carbamazepine, phenytoin, and barbiturates such as phenobarbital; strong inhibitors are HIV-antivirals, clarythromycin, itraconazole, ketoconazole, nefazodone, and telithromycin).
12. Incarcerated persons are excluded from the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-09-22 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Daver N, Cortes J, Newberry K, Jabbour E, Zhou L, Wang X, Pierce S, Kadia T, Sasaki K, Borthakur G, Ravandi F, Pemmaraju N, Kantarjian H, Verstovsek S. Ruxolitinib in combination with lenalidomide as therapy for patients with myelofibrosis. Haematologica. 2015 Aug;100(8):1058-63. doi: 10.3324/haematol.2015.126821. Epub 2015 Jun 18. PMID 26088933
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 2011- August 2013
Groups:
- Ruxolitinib + Lenalidomide: Ruxolitinib 15 mg orally twice daily continuously + Lenalidomide orally 5 mg/day on days 1-21, followed by 7 days of no therapy (28-day cycle). Prednisone will be added for patients who have not responded after 3 cycles of therapy. Prednisone 30 mg by mouth a day during cycle 4, 15 mg/day during cycle 5, and 15 mg every other day during cycle 6, and then it will be discontinued.
  Ruxolitinib: 15 mg by mouth twice daily (BID), continuously in 28-day cycles.
  Lenalidomide: 5 mg by mouth each day on days 1-21, followed by 7 days of no therapy of each 28 day cycle.
  Prednisone: Prednisone will be added for patients who have not responded after 3 cycles of therapy.
  30 mg by mouth a day during cycle 4, 15 mg/day during cycle 5, and 15 mg every other day during cycle 6, and then it will be discontinued.
Period: Overall Study
Arm/Group | Ruxolitinib + Lenalidomide
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib + Lenalidomide
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 17
Age, Continuous [Median (Full Range); unit: years] | 66 [37 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Participants With Objective Response
Description: To determine the efficacy of the combination of Ruxolitinib + Lenalidomide in patients with Myelofibrosis (MF). Objective response rate equals Complete and Partial Response, and Clinical Improvement as defined by International Working Group for Myelofibrosis Research and Treatment (IWG-MRT). Objective response rate (ORR), defined as a clinical improvement (CI), partial remission (PR), and complete remission (CR) according to the International Working Group (IWG) Criteria. Complete remission (CR): bone marrow blasts <5%, hemoglobin >/= 10, absolute neutrophil count (ANC) >/= 1000, platelets >/= 100, <2% immature myeloid cell, spleen and liver not palpable. Partial Response (PR): CR plus one or more of the following: ANC >/= 1000, decreased platelets by 50%, hemoglobin >/= 8.5 but < 10, <2% immature myeloid cells. Clinical improvement (CI): hemoglobin increase of 2g/dl, transfusion independence or reduction splenomegaly and/or hepatomegaly >/= 50%, >/=50% reduction in MPN-SAF TSS
Time Frame: 3 cycles (28 days each) up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib + Lenalidomide
Number analyzed (Participants) | 31
Participants | 7

ADVERSE EVENTS:
Time Frame: 6 years, 5 months
Arm/Group | Ruxolitinib + Lenalidomide
All-Cause Mortality (participants affected / at risk) | 2/31
Serious Adverse Events (participants affected / at risk) | 19/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib + Lenalidomide (N=31)
Neutropenic Fever (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Skin Infection (Infections and infestations) | 3 (9)
Lung Infection (Infections and infestations) | 8 (12)
Multi-Organ Failure (General disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superior Vena Cava Syndrome (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Chest pain (Cardiac disorders) | 1 (1)
Duodenal Infection (Infections and infestations) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Unspecified neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 1 (2)
Device related infection (Infections and infestations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Transient ischemic Attacks (Nervous system disorders) | 1 (2)
Death (General disorders) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib + Lenalidomide (N=31)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Ecchymosis-upper extremity (Blood and lymphatic system disorders) | 2 (2)
Edema limb (General disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 13 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (16)
Elevated ALT (Investigations) | 5 (5)
Elevated AST (Investigations) | 8 (8)
Hyperbilirubinemia (Investigations) | 5 (5)
Elevated Creatinine (Investigations) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Peripheral Neuropathy Motor (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT01375140/Prot_SAP_000.pdf